CLINICAL TRIAL: NCT05111223
Title: Testing the Contribution of Orbitofrontal Cortex Networks to Decision-making
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Christina Zelano, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00216104
Record Dates: First submitted 2021-10-28; First posted 2021-11-08 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMS targeting OFC anterior networks (Experimental): Participants will receive TMS and sham targeting the OFC network.
  Interventions: Device: Real transcranial magnetic stimulation (TMS) before conditioning; Device: Real transcranial magnetic stimulation (TMS) before devaluation test; Device: Sham transcranial magnetic stimulation (TMS)
- Experimental: TMS targeting posterior OFC networks (Experimental): Participants will receive TMS and sham targeting the posterior OFC network.
  Interventions: Device: Real transcranial magnetic stimulation (TMS) before conditioning; Device: Real transcranial magnetic stimulation (TMS) before devaluation test; Device: Sham transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Real transcranial magnetic stimulation (TMS) before conditioning — Real TMS will be applied using the MagVenture MagPro X100 stimulator with the active side of the Cool-B65 A/P coil before the conditioning phase of the task.
Device: Real transcranial magnetic stimulation (TMS) before devaluation test — Real TMS will be applied using the MagVenture MagPro X100 stimulator with the active side of the Cool-B65 A/P coil before the devaluation test phase of the task.
Device: Sham transcranial magnetic stimulation (TMS) — Sham TMS will be applied using the MagVenture MagPro X100 stimulator with the placebo side of the Cool-B65 A/P coil.

SUMMARY:
This research study examines the contribution of orbitofrontal cortex (OFC) networks to decision-making.

DETAILED DESCRIPTION:
This study will combine functional magnetic resonance imaging (fMRI), non-invasive transcranial magnetic stimulation (TMS), olfactory stimuli, and a devaluation task to define the specific contributions of orbitofrontal cortex (OFC) networks in outcome-guided behavior. We will use network-targeted TMS to modulate activity within anterior OFC and posterior OFC networks, examining if they have different contributions to decision-making. This is a randomized, between-subjects design.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years old
* Right-handed
* Fluent English speakers

Exclusion Criteria:

* History of significant neurological conditions (e.g., epilepsy, dementia, multiple sclerosis, brain tumors, etc.)
* History of major psychiatric conditions (e.g., general anxiety disorder, depression, schizophrenia, obsessive-compulsive disorder, post-traumatic stress disorder, attention deficit hyperactivity disorder, substance use disorder, etc.)
* Significant medical illnesses (e.g., cancer, meningitis, chronic obstructive pulmonary disease, cardiovascular disease, etc.)
* Significant cerebrovascular risk factors (e.g., hypertension, diabetes, elevated cholesterol, etc.)
* Current use of psychoactive medications (e.g., barbiturates, benzodiazepines, chloral hydrate, haloperidol, lithium, carbamazepine, phenytoin, citalopram, escitalopram, fluoxetine, diazepam, etc.)
* Smell or taste dysfunction
* History of significant allergies requiring hospitalization for treatment
* History of severe asthma requiring hospitalization for treatment
* Habitual smoking
* History of eating disorders (e.g., anorexia nervosa, bulimia nervosa, binge-eating disorder, etc.)
* Dieting or fasting
* Magnetic implants (e.g., shunts or stents, aneurysm clips, surgical clips, cochlear implants, metal bone/joint pins, plates and screws, eyelid spring or wires, etc.)
* Electronic devices (e.g., implanted cardiac defibrillator, cardiac pacemaker, deep brain/spinal cord or nerve stimulator, internal electrodes/wires, medication infusion devices, etc.)
* History of metal working without proper eye protection, or injury with metal shrapnel or metal slivers
* Claustrophobia
* Pregnancy
* Predisposition to seizures (e.g., personal history of seizures, family history of seizures epilepsy, pregnancy, alcoholism, etc.)
* Use of medications that increase the likelihood of seizures (e.g., bupropion SR, citalopram, duloxetine, ketamine, gamma-hydroxybutyrate, etc.)
* History of surgical procedures performed on the brain or spinal cord
* History of severe head trauma followed by loss of consciousness
* History of fainting spells or syncope
* Hearing problems or tinnitus

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Behavior on devaluation task | 1 hour after intervention
  Percentage of cues predicting non-devalued vs devalued odors chosen during the devaluation task.
Resting-state functional magnetic resonance imaging | 1 hour after intervention
  Resting-state activity determined by functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Zelano, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All data that underlie results in a publication
Time Frame: Upon publication
Access Criteria: Data can be obtained from PI for non-profit purposes upon reasonable request